CLINICAL TRIAL: NCT03115333
Title: Change in Relative Cerebral Blood Volume as a Biomarker for Early Response to Bevacizumab in Patients With Recurrent Glioblastoma
Brief Title: DSC-MRI in Measuring rCBV for Early Response to Bevacizumab in Patients With Recurrent Glioblastoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EAF151; NCI-2016-01357 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAF151 (Other: ECOG-ACRIN Cancer Research Group); EAF151 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2017-04-10; First posted 2017-04-14 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Gliosarcoma; Recurrent Glioblastoma
MeSH Terms: conditions — Gliosarcoma; Glioblastoma | interventions — Perfusion Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (DSC-MRI) (Experimental): Patients undergo DSC-MRI within 3 days before bevacizumab initiation and at day 15.
  Interventions: Diagnostic Test: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging — Undergo DSC-MRI
  Other Names: DSC-MRI; Dynamic Susceptibility Contrast-Enhanced MRI; DYNAMIC SUSCEPTIBILITY-CONTRAST MRI

SUMMARY:
This phase II trial studies how well dynamic susceptibility contrast-enhanced magnetic resonance imaging (DSC-MRI) works in measuring relative cerebral blood volume (rCBV) for early response to bevacizumab in patients with glioblastoma that has come back. DSC-MRI may help evaluate changes in the blood vessels within the cancer to determine a patient?s response to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether binary changes (increase versus [vs.] decrease) in rCBV within enhancing tumor from baseline to 2 weeks after initiation of anti-angiogenic therapy is associated with overall survival (OS).

SECONDARY OBJECTIVES:

I. To determine whether the baseline pre-treatment rCBV measure alone is associated with OS.

II. To determine whether binary changes (increase vs. decrease) in rCBV within enhancing tumor from baseline to 2 weeks after initiation of anti-angiogenic therapy is associated with progression-free survival (PFS).

III. To determine whether changes in rCBV as a continuous variable within enhancing tumor from baseline to 2 weeks after initiation of anti-angiogenic therapy is associated with OS or PFS.

IV. To determine the association between rCBV and OS when adjusting for the changes in enhancing tumor volume.

V. To determine whether baseline cerebral blood flow (CBF) or change in CBF is associated with OS or PFS.

OUTLINE:

Patients undergo DSC-MRI within 3 days before bevacizumab initiation and at day 15.

After completion of study intervention, patients are followed up every 3 months for 1 year and then every 6 months for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven intracranial glioblastoma or gliosarcoma at initial surgery

  * Patients will be eligible if the original histology was low-grade glioma and a subsequent diagnosis of glioblastoma or gliosarcoma is made (high-grade transformation)
* Karnofsky performance status >= 70
* Women must not be pregnant or breast-feeding
* Progression of disease assessed by local site using Revised Assessment in Neuro-Oncology (RANO) criteria, with plan to give whole-dose bevacizumab therapeutically, either as single therapy or in conjunction with other chemotherapeutic regimens; patients getting bevacizumab to support additional radiation therapy or immunotherapy, or primarily for reduction of edema rather than for tumor treatment, are excluded; this must be the patient?s initial recurrence
* Patient must not have been treated previously with immunotherapies (vaccines, checkpoint inhibitors, T-cells)
* Intratumoral hemorrhage (acute, subacute, or chronic) as seen on hemosiderin-sensitive (gradient-echo) MRI may preclude patient inclusion because of anticipated limited evaluation due to magnetic susceptibility artifact on the heavily T2-weighted DSC-MRI images; if the region of enhancing tumor not affected by blooming artifact on the hemosiderin-sensitive images does not meet the 10 x 10 x 10 mm ?measurable enhancement? threshold specified elsewhere, the patient is ineligible
* Progressive enhancement (> 25% increase in contrast enhancing volume compared to nadir) on MRI within 14 days of registration, >= 42 days since completion of radiation/temozolomide therapy, and >= 28 days since surgical resection or cytotoxic chemotherapy; measurable enhancement is defined as two perpendicular in-plane diameters of at least 10 mm and at least 10 mm in the 3rd orthogonal direction
* Patients must be able to tolerate brain MRI scans with dynamic intravenous gadolinium-based contrast agent injections

  * Ability to withstand 22 gauge intravenous (IV) placement
  * No history of untreatable claustrophobia
  * No magnetic resonance (MR) incompatible implants/devices or metallic foreign bodies
  * No contraindication to intravenous contrast administration

    * Adequate organ function, including adequate renal function defined as estimated glomerular filtration rate (eGFR) >= 40 mL/min/1.73 m^2 as calculated per institution standard of care, and meeting local site requirements for intravenous administration of gadolinium-based MRI contrast agents
  * No known allergy-like reaction to gadolinium or moderate or severe allergic reactions to one or more allergens as defined by the American College of Radiology (ACR); patient may be eligible if willing to undergo pre-treatment as defined by the institution's policy and/or ACR guidance
  * Weight compatible with limits imposed by the MRI scanner table
* Patient must be scheduled to receive treatment with a standard dose regimen of bevacizumab (bevacizumab infusion on days 1 and 15 of a 28-day treatment cycle); patient can be treated with bevacizumab alone or in combination with other chemotherapies Exclusion Criteria: (see Inclusion Criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2027-05-07 (Estimated)

PRIMARY OUTCOMES:
Change in rCBV within enhancing tumor | Baseline to 2 weeks
  Will determine whether binary changes (increase vs. decrease) in rCBV is associated with OS. Kaplan-Meier survival curves will be generated for both the increased and the decreased rCBV groups. The median survival time of both groups will be estimated and compared with a two-sided log rank test. Univariate Cox proportional hazards model will be used to test the association between changes in rCBV from baseline to 2 weeks and OS or PFS.
OS | Up to 5 years
  Will determine if binary changes (increase vs. decrease) in rCBV is associated with OS. The median survival time of both groups will be estimated and compared with a two-sided log rank test. Will determine whether changes in rCBV as a continuous variable within enhancing tumor from baseline to 2 weeks after initiation of anti-angiogenic therapy is associated with OS. Univariate Cox proportional hazards model will be used to test the association between changes in rCBV from baseline to 2 weeks and OS. The hazard ratio and its 95% confidence interval (CI) will be presented. Will determine the as

SECONDARY OUTCOMES:
CBF | Baseline
  Will determine if baseline CBF is associated with OS or PFS. Kaplan-Meier survival curves will be generated for both the increased and the decreased CBF groups, for either OS or PFS. The median survival time/progression free survival time of both groups will be estimated and compared with a two-sided log rank test. Univariate Cox proportional hazards model will be used to test the association between baseline CBF and OS or PFS. The hazard ratio and its 95% CI will be presented.
Change in CBF | Baseline to 2 weeks
  Will determine if changes in CBF is associated with OS or PFS. Kaplan-Meier survival curves will be generated for both the increased and the decreased CBF groups, for either OS or PFS. The median survival time/progression free survival time of both groups will be estimated and compared with a two-sided log rank test. The hazard ratio and its 95% CI will be presented.
PFS | Up to 5 years
  Will determine whether binary changes (increase vs. decrease) in rCBV within enhancing tumor from baseline to 2 weeks after initiation of anti-angiogenic therapy is associated with PFS. Will determine whether changes in rCBV as a continuous variable within enhancing tumor from baseline to 2 weeks after initiation of anti-angiogenic therapy is associated with PFS. Univariate Cox proportional hazards model will be used to test the association between changes in rCBV from baseline to 2 weeks and PFS. Kaplan-Meier survival curves will be generated for both the increased and the decreased rCBV grou
rCBV | Baseline
  Will determine whether the baseline pre-treatment rCBV measure alone is associated with OS. Univariate Cox proportional hazards model will be used to test the association between baseline rCBV and OS. The hazard ratio and its 95% confidence interval will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Boxerman, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (58):
- United States (58):
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Eden Hospital Medical Center, Castro Valley, California
  - Loma Linda University Medical Center, Loma Linda, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, East White Plains, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin